CLINICAL TRIAL: NCT06316908
Title: Permanent Celiac Plexus Block: Comparison of Pain Score in Unilateral and Bilateral Posterior Percutaneous Approach
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sindh Institute of Urology and Transplantation (Other)
Responsible Party: Principal Investigator, Syed Muhammad Abbas, Associate Professor, Department of Anaesthesia, Sindh Institute of Urology and Transplantation
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ERC-2019/A187
Record Dates: First submitted 2024-01-21; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Abdominal Cancer; Cancer Pain; Cancer of Pancreas
MeSH Terms: conditions — Cancer Pain; Pancreatic Neoplasms | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Unilateral Approach Group: Patients in this group have received a unilateral percutaneous posterior approach for NCPB. The procedure was performed under fluoroscopic guidance.
  Bilateral Approach Group: Patients in this group have undergone a bilateral percutaneous posterior approach for NCPB, following the same procedural guidance.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Unilateral Approach Group (Active Comparator): Patients in this group have received a unilateral percutaneous posterior approach for NCPB. The procedure was performed under fluoroscopic guidance
  Interventions: Drug: Unilateral Neurolytic Celiac Plexus Block with Absolute Alcohol
- Bilateral Approach Group (Active Comparator): Patients in this group have undergone a bilateral percutaneous posterior approach for NCPB, following the same procedural guidance.
  Interventions: Drug: Bilateral Neurolytic Celiac Plexus Block with Absolute Alcohol

INTERVENTIONS:
Drug: Unilateral Neurolytic Celiac Plexus Block with Absolute Alcohol — Participants assigned to the unilateral neurolytic celiac plexus block group underwent a minimally invasive procedure where a solution of absolute alcohol was injected unilaterally into the celiac plexus under image guidance. The procedure was performed by an experienced interventional pain specialist. Prior to the injection, local anesthesia was administered to minimize discomfort. Once positioned correctly, a needle was inserted into the designated area, and a small amount of absolute alcohol was injected to disrupt the neural pathways responsible for transmitting pain signals from the abdominal region. The intervention aims to provide long-term pain relief for participants suffering from chronic abdominal pain.
  Arms: Unilateral Approach Group
Drug: Bilateral Neurolytic Celiac Plexus Block with Absolute Alcohol — Participants allocated to the bilateral neurolytic celiac plexus block group underwent a similar minimally invasive procedure as described above, with the exception that the injection of absolute alcohol was administered bilaterally into the celiac plexus. The procedure was performed by an experienced interventional pain specialist under image guidance, with local anesthesia administered prior to the injection to ensure patient comfort. Following correct needle placement, absolute alcohol was injected into both sides of the celiac plexus to disrupt neural pathways responsible for transmitting pain signals from the abdominal region. The intervention aims to provide comparable or potentially enhanced long-term pain relief compared to the unilateral approach, with the additional benefit of targeting both sides of the celiac plexus.
  Arms: Bilateral Approach Group

SUMMARY:
The goal of this prospective, interventional, non-randomized study was to compare pain score in unilateral and bilateral posterior percutaneous neurolytic celiac plexus block (NCPB) in upper abdominal cancer patients.

The main questions it aimed to answer are:

1. Whether unilateral or bilateral NCPB technique has a better pain relief
2. Was there any difference in terms of complication rates between these two approaches All participants were having upper abdominal cancer whether operated or non-operable cancer were given a unilateral or bilateral neurolytic celiac plexus block.

Pain scores and adverse events at multiple time points post-procedure were recorded.

DETAILED DESCRIPTION:
After Institutional Research Committee clearance and Ethical Review Committee approval from the Sindh Institute of Urology & Transplantation, the patients were divided into two groups, 15 patients in each group. Forty milliliters of the study drug were prepared in a 50 milliliters (mL) syringe by a pharmacy person. Patients were nil per oral (NPO) for six hours and after a written informed consent, patients were brought in the operating room. A 20-gauge (G) intravenous (I/V) cannula was passed and started injection ringer lactate at 10 mL/kg body weight, for all patients except diabetic mellitus who received normal saline. Monitors were applied as per American Society of Anesthesiologist (ASA) standards i.e., electrocardiogram (ECG), oxygen saturation (SpO2), and non-invasive blood pressure (NIBP), and vitals were recorded at intervals of 5 minutes (min). Patients were then positioned prone on the operation table and their arms were rested on the arm board. Pillows were placed under the abdomen between the ribs and iliac crest.

First, a mark was made between the 12 Thoracic (T12) and 1st Lumbar (L1) vertebra under the Fluoroscopic C arm view. Then a line was drawn between the points at 5 and 7 cm lateral from the spinous process of the L3 vertebra. Injection 2% plain xylocaine 3-5 milliliters (mL) was locally infiltrated and a 20-centimeter (cm) 22gauge (G) Chiba needle was inserted at an angle of 45 degrees with the skin and directed medially and in cephalic direction. After making contact with the body of the L1 vertebra needle was withdrawn and reinserted with an increased angle between the needle shaft and the skin until the tip of the needle slipped off the body of the L1 vertebra. Then the needle was advanced 1-1.5 cm in front of the T12 & L1 vertebrae. The position of the needle was confirmed in the anterior and lateral views of the vertebra with the help of radiopaque dye under a fluoroscopic C arm view. After the proper confirmation of the tip of the needle, 40 mL of absolute alcohol was injected into the unilateral block. Whereas, in the bilateral technique 20 mL absolute alcohol on both sides were injected. During and after the drug administration the pattern of the drug distribution was observed very carefully anterior to the body of the L1 vertebra and psoas fascia, and any visceral and I/V drug administration was avoided. After alcohol administration, 0.25 % Bupivacaine 5 mL was given, and then withdrawn the needle. The patient remained in the prone position for 20 mins. After the patients were turned supine and shifted to the post-anesthesia care unit (PACU) for monitoring of vitals for 30 mins after which they shifted to the ward. Pain score was recorded immediately and then at 30 mins in PACU, then at 6, 12, and 24 hours. Patients were discharged after 24 hours or when stable, pain score was recorded on telephonic conversation/ outpatient clinic visits at 7 days, 1 month, 3 months, and 6 months after the procedure or till death if the patient expired before 6 months.

ELIGIBILITY:
Inclusion Criteria:

* All upper abdominal malignancy adult patients
* on palliative care,
* having a visual analog scale (VAS) of more than 7

Exclusion Criteria:

* Patients on anti-coagulant medications,
* having an INR > 1.50 and or
* Platelets count < 80000,
* inability to provide informed consent, or
* those who have previously undergone celiac plexus intervention.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Pain Score using the Visual Analog Scale | 6 months post-procedure
  The visual analog scale consists of a 10 cm long horizontal line, with a minimum value of 0 (no pain) and a maximum value of 10 (worst pain imaginable). Higher scores indicate a worse outcome.

SECONDARY OUTCOMES:
Change in Mean Arterial Pressure | 4 hours post-procedure
  Change in mean arterial pressure from baseline (pre-procedure) to 4 hours post-procedure. Mean arterial pressure was measured by a non-invasive automated blood pressure reader.
Incidence of Patient-Reported Nausea Feeling | 24 hours post-procedure
  Nausea was defined as patient reported feeling of urge to vomit. The incidence will be reported as the percentage of patients who report experiencing nausea at least once during the follow-up period.
Incidence of Vomiting | 24 hours post-procedure
  The occurrence and frequency of vomiting was documented through patient self-reporting or clinical observation.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Q Abbas, MCPS, FCPS, Principal Investigator — Professor Dept of Anaesthesia
Locations (1):
- Sindh Institute of Urology and Transplantation, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No